CLINICAL TRIAL: NCT01443884
Title: Anti-Inflammatory Activities of Grapes in Humans at Risk for Cardiovascular Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: USDA, Western Human Nutrition Research Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 200816801-2
Record Dates: First submitted 2011-09-28; First posted 2011-09-30 (Estimated); Last update posted 2011-12-12 (Estimated); Status verified 2011-12

CONDITIONS: Obesity; Inflammation
MeSH Terms: conditions — Obesity; Inflammation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Experimental): After a 1 week baseline, volunteers will consume two packets of grape powder stirred into water for three weeks. Each packet will contain the equivalent of approximately 2 servings of fresh grapes (46 grams of powder). Following a two week washout period, volunteers will cross-over to a placebo powder.
  Interventions: Dietary Supplement: Grape powder, followed by placebo powder
- Group 2 (Experimental): After a 1 week baseline, volunteers will consume two packets of placebo powder stirred into water for three weeks. Following a two week washout period, volunteers will cross-over to grape powder for three weeks.
  Interventions: Dietary Supplement: Placebo powder followed by grape powder

INTERVENTIONS:
Dietary Supplement: Grape powder, followed by placebo powder — For three weeks, twice per day, volunteers will consume one packet of freeze-dried grape powder containing the equivalent of approximately 2 servings of fresh grapes (46 grams of powder) stirred into water. Following a two week washout, volunteers will consume one packet of placebo powder twice per day for three weeks.
  Arms: Group 1
Dietary Supplement: Placebo powder followed by grape powder — For three weeks, twice per day, volunteers will consume one packet of placebo powder stirred into water. Following a two week washout, volunteers will consume one packet of freeze-dried grape powder containing the equivalent of approximately 2 servings of fresh grapes (46 grams of powder) twice per day for three weeks.
  Arms: Group 2

SUMMARY:
The goal of the study is to determine whether grape consumption can reduce the risk of cardiovascular disease by reducing the presence of inflammatory molecules and positively altering cholesterol levels, lipid profiles, and immune cell responses.

DETAILED DESCRIPTION:
Obese individuals are at high risk for the development of hypertension and cardiovascular disease. Adipose tissue is a major source of pro-inflammatory molecules which can promote the development of atherosclerosis. Development of atherosclerotic plaques are mediated by oxidized or otherwise modified LDL cholesterol and infiltration of activated immune cells into the atherosclerotic lesions. Grapes contain high levels of polyphenols, a class of compounds known to possess antioxidant and anti-inflammatory properties. The overall goal of this proposal is to determine whether grape consumption can reduce the risk of cardiovascular disease by reducing the presence of inflammatory molecules and positively altering cholesterol levels, lipid profiles, and immune cell responses. Using a randomized cross-over design, twenty obese subjects will consume beverages containing either four servings of grape powder per day or the caloric equivalent without grape powder (placebo control) for a total of three weeks. After a two week washout period, the beverages will be switched for a further three weeks. Blood will be taken from each person at six intervals to determine lipid profiles, measure inflammatory markers in plasma, and analyze immune cell responsiveness.

ELIGIBILITY:
Inclusion Criteria:

* BMI 30 - 45 kg/m2
* Commitment to the dietary intervention and scheduled testing

Exclusion Criteria:

* Subjects will be excluded from this study if their blood cell counts or blood chemistry profiles are outside of the normal range
* smoking or use of tobacco products
* drink more than one alcoholic beverage per day (1 oz. distilled liquor, 3 oz. wine, or 12 oz. beer)
* taking cholesterol-lowering medications
* taking steroids for asthma or other inflammatory states
* taking thyroid-regulating drugs
* taking over-the counter weight loss products

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2009-10; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Change in inflammatory mediators in serum | 0, 1, 3, 4, 8, and 9 weeks
  C-reactive protein, serum amyloid A, cytokines (IL-1, IL-6, IL-8, and TNF-a), and soluble adhesion molecules (sICAM-1, sVCAM-1) will be measured.

SECONDARY OUTCOMES:
Change in lipid particle size and quantity | 0, 1, 3, 4, 8 and 9 weeks
  Lipid particle size will be measured using NMR spectroscopy, inlcuding chylomicrons, six VLDL subpopulations, IDL, three LDL subpopulations, and five HDL subpopulations.
CHange in activation and proliferation of T lymphocytes | 0, 1, 3, 4, 8 and 9 weeks
  Activation and proliferative responses of T lymphocytes will be measured to determine if grape consumption alters immune cell responsiveness. Proliferative responses will be measured using flow cytometry.

CONTACTS AND LOCATIONS:
Overall Officials: Susan Zunino, PhD, Principal Investigator — USDA, ARS, Western Human Nutrition Research Center
Locations (1):
- USDA, ARS, Western Human Nutrition Research Center, Davis, California, United States